CLINICAL TRIAL: NCT01783912
Title: Preparing Those With Significant and Persistent Mental Illness to Quit Smoking
Brief Title: Helping Those With Mental Illness Quit Smoking
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-0604
Record Dates: First submitted 2013-01-22; First posted 2013-02-05 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Smoking; Nicotine Dependence; Mental Disorders
Keywords: Smoking; Nicotine Dependence; Mental Disorders
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Mental Disorders | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cognitive/Motivational Intervention Group (Experimental): This arm of the project will address the following questions:
  After completion of experimental individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Active Control group?
  After completion of experimental individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Motivated Smokers Comparison group?
  Interventions: Behavioral: Cognitive / Motivational Individual Sessions; Drug: Nicotine Patch; Behavioral: Group Curriculum
- Attention Control Group (Active Comparator): This arm of the project will address the following question:
  After completion of control individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate that those who are in the experimental treatment group?
  After completion of control individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Cognitive/Motivational Intervention Group?
  Interventions: Behavioral: Attention Control Individual Sessions; Behavioral: Group Curriculum
- Motivated Smokers Comparison Group (No Intervention): This arm of the project will address the following question:
  Do participants in the Motivated Smokers Comparison group (identified as motivated to quit upon recruitment) utilize the quit line services at the same, greater or lesser rate than those who are in the Motivated Smokers Comparison group?
  Do participants in the Motivated Smokers Comparison group (identified as motivated to quit upon recruitment) utilize the quit line services at the same, greater or lesser rate than those who are in the Active Control group?
  Participants will not receive any intervention but will be consented and enrolled into this group and assessed for utilization of the tobacco quit line services.

INTERVENTIONS:
Behavioral: Cognitive / Motivational Individual Sessions — Cognitive Motivational subjects will receive four evidence-based preparatory interventions (motivational interviewing, smoking reduction, practice quit attempt, and pre-quit use of nicotine replacement medication) (25 - 30 minutes each).
  Arms: Cognitive/Motivational Intervention Group
Behavioral: Attention Control Individual Sessions — Attention control subjects will receive four placebo individual sessions (25-30 minutes each). The session content will reemphasize group discussion of the personal health risks from smoking.
  Arms: Attention Control Group
Drug: Nicotine Patch — Cognitive Motivational subjects will be asked to take one 21 mg patch/day for 4 weeks.
  Arms: Cognitive/Motivational Intervention Group
Behavioral: Group Curriculum — Everyone to be put into the experimental or active comparator group will attend 2 group meetings over two weeks each of which lasts 40 minutes. Experience with the Kicking Butts program indicates that this duration is well tolerated by this population. The content of these two group meetings is based on the Kicking Butts program. The Kicking Butts program was initially developed as a cessation intervention, but consistent with the literature about the need to prepare this population to make a quit attempt, has evolved to emphasize preparation for quitting. Topics addressed include the health consequences of smoking, reasons to quit and methods of quitting.
  Arms: Attention Control Group; Cognitive/Motivational Intervention Group

SUMMARY:
This study tests whether pre-cessation interventions known to be effective in the general population will increase acceptance of evidence-based treatment, engagement and compliance with that treatment and initial quitting success. One hundred and seventy two patients will be recruited from 13 Community Support Programs (CSPs). CSPs provide community based care to those diagnosed with persistent and serious mental illness. All participants will receive two group sessions (40 minutes each) modeled after "Kicking Butts", a group-based quitting preparation program used for the past four years in two Milwaukee CSP programs run by Wisconsin Community Services. Individuals will then be randomly assigned to the experimental and control conditions (n=86 each). Experimental subjects will receive four evidence-based preparatory interventions (motivational interviewing, smoking reduction, practice quit attempt, and pre-quit use of nicotine replacement medication) (25 - 30 minutes each). Attention control subjects will also receive four individual sessions of the same duration. However their individual sessions' content will be a discussion of the personal relevance of the group material and will not include any of the preparatory interventions. Data will be collected via brief surveys taken pre-intervention, at the end of the last individual session, and three months later and from a database provided by the Wisconsin Tobacco Quit Line (WTQL).

ELIGIBILITY:
Inclusion Criteria:

* current smoker (smoking daily or smoking at least 10 cigarettes per week) (use of other tobacco products permitted such as chew and snuz in addition to smoking)
* not willing to make a quit attempt
* willingness to use the nicotine patch
* plans to remain in the area for the next five four months.

Exclusion Criteria:

* current use of any cessation medicine (nicotine patch, nicotine gum, nicotine lozenge, nicotine inhaler, nicotine nasal spray, bupropion, Wellbutrin, Zyban,Chantix or varenicline)
* previous serious skin reaction or other allergic reaction to using the nicotine patch
* stroke, heart attack or abnormal electrocardiogram in past four weeks
* pregnancy, plans to get pregnant or nursing
* exclusive use of other tobacco products (non-smoker tobacco user)
* having a court-ordered guardian, or an activated power of attorney for health or observation by researchers during the consent procedure that suggests diminished decision making capacity

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Christiansen, PhD, Principal Investigator — University of Wisconsin School of Medicine and Public Health, Center for Tobacco Research and Intervention
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin School of Medicine and Public Health, Center for Tobacco Research and Intervention Website — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitive/Motivational Intervention Group: This arm of the project will address the following questions:
  After completion of experimental individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Active Control group?
  After completion of experimental individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Motivated Smokers Comparison group?
  Cognitive / Motivational Individual Sessions: Cognitive Motivational subjects will receive four evidence-based preparatory interventions (motivational interviewing, smoking reduction, practice quit attempt, and pre-quit use of nicotine replacement medication) (25 - 30 minutes each).
  Nicotine Patch: Cognitive Motivational subjects will be asked to take one 21 mg patch/day for 4 weeks.
- Attention Control Group: This arm of the project will address the following question:
  After completion of control individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate that those who are in the experimental treatment group?
  After completion of control individual sessions, do the participants in the control group utilize the quit line services at the same, greater or lesser rate than those who are in the Cognitive/Motivational Intervention Group?
  Attention Control Individual Sessions: Attention control subjects will receive four placebo individual sessions (25-30 minutes each). The session content will reemphasize group discussion of the personal health risks from smoking.
Period: Overall Study
Arm/Group | Cognitive/Motivational Intervention Group | Attention Control Group | Motivated Smokers Comparison Group
Started | 118 | 104 | 48
Completed | 88 | 58 | 25
Not Completed | 30 | 46 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive/Motivational Intervention Group | Attention Control Group | Motivated Smokers Comparison Group | Total
Number analyzed (Participants) | 118 | 104 | 48 | 270
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.88) | 43.6 (10.05) | 45.0 (9.54) | 44.0 (9.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 48 | 24 | 130
  Male | 60 | 56 | 24 | 140
Region of Enrollment [Number; unit: participants]
  United States | 118 | 104 | 48 | 270

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of Wisconsin Tobacco Quit Line Services
Description: The primary outcome is participant acceptance of evidence based treatment through the WTQL at the end of the last individual session.
Time Frame: 4-6 weeks after study enrollment
Measure: Number; unit: participants
Arm/Group | Cognitive/Motivational Intervention Group | Attention Control Group | Motivated Smokers Comparison Group
Number analyzed (Participants) | 118 | 104 | 48
participants | 11 | 6 | 6

ADVERSE EVENTS:
Arm/Group | Cognitive/Motivational Intervention Group | Attention Control Group | Motivated Smokers Comparison Group
Serious Adverse Events (participants affected / at risk) | 0/118 | 0/104 | 0/48
Other Adverse Events (participants affected / at risk) | 0/118 | 0/104 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No